CLINICAL TRIAL: NCT05708261
Title: Tailoring Healthy Relationships to Improve HIV Outcomes for MSM in Eastern Cape, South Africa
Brief Title: Tailoring Healthy Relationships to Improve HIV Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Foundation for Professional Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00014539
Record Dates: First submitted 2022-02-18; First posted 2023-02-01 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: HIV

STUDY DESIGN:
Intervention Model Description: This is a behavioral intervention designed to provide HIV communication and disclosure skill building to improve treatment adherence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MR Intervention (Experimental): Grounded in Social Cognitive Theory, the intervention delivers five 2-hour sessions with 3 post-session group check-in's to develop skills in partnership communication, HIV disclosure and prevention. The intervention utilizes self-assessments on skills learned and then action plan for these developed and then finalized in the last session.
  Interventions: Behavioral: MR Intervention
- Be Well (Other): Attention match control arm. Participants will receive standard of care for HIV treatment and one-way SMS with video content about general health. This will occur once per week during the first 5 weeks after enrollment.
  Interventions: Other: Be Well Attention Match

INTERVENTIONS:
Behavioral: MR Intervention — Grounded in Social Cognitive Theory, the intervention delivers five 2-hour sessions with 3 post-session group check-in's to develop skills in partnership communication, HIV disclosure and prevention. The intervention utilizes self-assessments on skills learned and then action plan for these developed and then finalized in the last session.
  Arms: MR Intervention
Other: Be Well Attention Match — Attention match control arm providing one-way SMS of general health content delivered once per week during the first 5 weeks after enrollment.
  Arms: Be Well

SUMMARY:
This study will adapt the evidence-based intervention, Healthy Relationships, and then assess its feasibility using a pilot randomized controlled trial with HIV-positive MSM living with HIV in Eastern Cape, South Africa

DETAILED DESCRIPTION:
This project will adapt the intervention, Healthy Relationships (HR), and then conduct a pilot test of the intervention in Eastern Cape, South Africa, with HIV positive men who have sex with men (MSM). HR is a group based intervention designed to develop participant skills in assessing HIV stress and communication skills for disclosure and safe sex. This original intervention was developed with MSM and subsequently adapted for video conference (VC) delivery with women in the U.S. The adaptation will include updated HIV education and focus on MSM in relationship because limited HIV disclosure and prevention risk assessment and communication skills are associated with lowered ART adherence, and the intervention will be named MPowered in Relationships (MR). Similar to the VC version of HR for women, investigators will deliver MR via Zoom followed by three group check ins via Zoom as well. The check ins will review MR skills learned and applied including assessing individual action plans in these areas. Also, through this project, investigators will develop a community advisory board that will guide intervention adaptation. The outcomes of the pilot-test are to assess feasibility, acceptability, willingness and safety of the MR, as well as assess the potential impact of the intervention on behavioral measures, ART adherence and viral load. Our hypothesis is that HIV disclosure and prevention skill will be feasible and demonstrate a preliminary impact on behavioral and biomedical measures that will support a clinical trial of the intervention.

After adaptation of the intervention, Healthy Relationships (HR), with enhanced components for MSM (Aim 1) and then a pilot test of the intervention to determine if it is feasible in Eastern Cape, South Africa (Aim 2). The name of this intervention will be MR. The proposed project is based on preliminary research conducted by the principal investigators, and the study is benefitting from collaborations with the Foundation for Professional Development in Eastern Cape, South Africa.

Intervention adaptation (Aim 1) will use mixed methods to include interviews with MSM and health experts to integrate updated HIV prevention and treatment education (PrEP, U=U) and contextual components to ensure skill-building for HIV communication and disclosure risk assessment. This aim will include a usability test to ensure conceptual understanding of the intervention content by MSM to finalize adaptation. This feasibility study (Aim 2) will be a pilot-test using a randomized controlled trial design.

In Specific Aim 2, investigators will pilot test the adapted intervention, MR, with HIV positive MSM in Eastern Cape, South Africa. The outcomes for this pilot are to understand feasibility (feasibility, acceptability, willingness, and safety) and preliminary impact on behavioral and biomedical outcomes of the intervention for this group. The findings from this pilot study will be used to inform a larger clinical trial to determine the effectiveness of MR in reducing HIV disclosure, prevention and treatment outcomes for MSM in this setting. The pilot study will be a randomized controlled trail with participant recruited from MSM specific HIV activities in Eastern Cape, and then investigators will be randomly assigned to either the intervention or control groups. The study design will include an attention matched control in order to reduce the effect of other mHealth tools that MSM may be experiencing during the study. The intervention will complete MR, and the attention matched control arm will complete Be Well.

MR: One MR session will be delivered per week for five weeks over Zoom, and then three group check ins will be conducted eight, twelve and sixteen weeks. Each of the original five HR sessions will be divided into two one hour sessions and delivered via Zoom where participants will access using their personal smartphone. During the intervention, participants will complete viral load tests at baseline and post intervention. Also, participants will complete behavioral assessments at baseline, mid study, post intervention, and follow up at 16 months. For baseline and post intervention, the behavioral assessment will measure areas like HIV treatment knowledge, internalized HIV stigma, HIV care self efficacy, alcohol use, HIV disclosure, safe sex practices, relationship factors, and ART adherence behaviors. In addition, each participant will complete MR feasibility interview during study visit with a feasibility survey that will be completed at post intervention.

Be Well: The attention matched control arm will involve general health video links sent via SMS to participant smartphones and one way, informational SMS on general health and wellness that are not HIV related. The videos and SMS content will be based on the BWise online website that is run by the Ministry of Health in South Africa. The attention matched control participants will complete the same viral load and behavioral measures as the intervention arm, but participants will not complete the MR feasibility interview and survey.

Data Analysis: Qualitative interview data will be analyzed using a constant comparison approach, with comparisons by age, sexuality, HIV diagnosis date, and time of interview (baseline, mid, post intervention) in the themes identified. Investigators will analyze the feasibility survey and MR paradata (CommCare and Zoom) using univariate statistics and compare prevalence/mean (range) by age, sexuality, HIV diagnosis date, and study group using appropriate statistical tests for significance. For the behavioral outcomes, investigators will examine univariate properties (frequency and range) and compare prevalence/mean (range) by age, sexuality, HIV diagnosis date, and study group using appropriate statistical tests for significance. Investigators will conduct additional analysis of the prevalences and means (ranges) of these variables across the intervention and attention matched arms, focusing on identifying significant differences in changes in these variables pre and post intervention. For viral load, since there is limited knowledge on the effects of interventions on viral load for MSM in this setting, investigators will examine univariate properties (frequency and range) of viral load within each arm and compare prevalence mean (range) by age, sexuality, HIV diagnosis date, study group, and ART adherence patterns. Undetectable HIV viral load (fewer than 50 copies of HIV per millimeter of blood) will not be an expected outcome for this study, but the analysis will provide viral load range to inform a larger clinical trial.

ELIGIBILITY:
INCLUSION CRITERIA:

Aim 1 MSM

1. 18 years of age or older
2. MSM by self-report
3. HIV-positive status confirmed by HIV self-test
4. Sub-optimal ART adherence confirmed by Visual Analog Scale
5. Live in Eastern Cape confirmed by map exercise
6. Mentally competent to provide voluntary informed consent
7. Prescribed ART
8. Own a smartphone for personal use
9. Comfortable talking about living with HIV and relationships in group settings
10. In a relationship with a man (defined as a boyfriend, partner, husband, lover) with whom they are emotionally and romantically connected to all others.
11. Have not disclosed HIV-positive status to partner
12. Partner status is unknown or HIV-negative

Health Professional and Technical Experts

1. Provide clinical care (medical or nursing) to MSM in Eastern Cape, South Africa (Health Professionals only)
2. Experience developing mobile technologies for HIV prevention and treatment in Eastern Cape, South Africa (Technical Experts only)
3. Live in Eastern Cape, South Africa
4. Mentally competent to provide voluntary informed consent

Community Advisory Board

1. Identifies as MSM
2. In a relationship with a man
3. Participates in HIV-related activities focused on MSM
4. 18-25 years of age (N=4) or 26 years of age and older (N=4)
5. Lives in Eastern Cape

Aim 2 MSM (only)

1. 18 years of age or older
2. MSM by self-report
3. HIV-positive status confirmed by HIV self-test
4. Sub-optimal ART adherence confirmed by Visual Analog Scale
5. Live in Eastern Cape confirmed by map exercise
6. Mentally competent to provide voluntary informed consent
7. Prescribed ART
8. Own a smartphone for personal use
9. Comfortable talking about living with HIV and relationships in group settings
10. In a relationship with a man (defined as a boyfriend, partner, husband, lover) with whom they are emotionally and romantically connected to all others and the relationship is more than 1 month old.
11. Have not disclosed HIV-positive status to partner
12. Partner HIV-status is unknown or HIV-negative

EXCLUSION CRITERIA:

Aim 1 MSM

1. Under 18 years of age
2. Is not MSM by self-report
3. Is not HIV-positive as confirmed by HIV self-test
4. Does not have sub-optimal ART adherence confirmed by Visual Analog Scale
5. Does not live in Eastern Cape confirmed by map exercise
6. Is not mentally competent to provide voluntary informed consent
7. Not prescribed ART
8. Does not own a smartphone for personal use
9. Is not comfortable talking about living with HIV and relationships in group settings
10. Not in a relationship with a man (defined as a boyfriend, partner, husband, lover) with whom they are emotionally and romantically connected to all others or in this defined relationship for less than a month.
11. Has disclosed their HIV-positive status to partner
12. Partner is HIV-positive

Health Professional and Technical Experts

1. Does not provide clinical care (medical or nursing) to MSM in Eastern Cape, South Africa (Health Professionals only)
2. No experience developing mobile technologies for HIV prevention and treatment in South Africa (Technical Experts only)
3. Does not live in Eastern Cape, South Africa
4. Not mentally competent to provide voluntary informed consent

Community Advisory Board

1. Does not identify as MSM
2. Is not in a relationship with a man
3. Does not participate in HIV-related activities focused on MSM
4. Is not 18-25 years of age (N=4) or 26 years of age and older (N=4)
5. Does not live in Eastern Cape

Aim 2 MSM (only)

1. Under 18 years of age
2. Is not MSM by self-report
3. Is not HIV-positive as confirmed by HIV self-test
4. Does not have sub-optimal ART adherence confirmed by Visual Analog Scale
5. Does not live in Eastern Cape confirmed by map exercise
6. Is not mentally competent to provide voluntary informed consent
7. Not prescribed ART
8. Does not own a smartphone for personal use
9. Is not comfortable talking about living with HIV and relationships in group settings
10. Not in a relationship with a man (defined as a boyfriend, partner, husband, lover) with whom they are emotionally and romantically connected to all others, or in this defined relationship for less than a month.
11. Has disclosed their HIV-positive status to partner
12. Partner is HIV-positive

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-29 (Estimated); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
Feasibility Survey | Month 3
  A study specific survey to assess feasibility, willingness, safety, acceptability
Feasibility Survey | Month 6
  A study specific survey to assess feasibility, willingness, safety, acceptability
Feasibility Interview | Month 3
  Indepth interview to assess feasibility, willingness, safety, acceptability
Feasibility Interview | Month 6
  Indepth interview to assess feasibility, willingness, safety, acceptability

SECONDARY OUTCOMES:
HIV viral load | Month 0
  Collect Dried Blood Spots to measure for viral load
HIV viral load | Month 9
  Collect Dried Blood Spots to measure for viral load
HIV treatment adherence | Month 0
  A survey to assess dosing of antiretroviral medication
HIV treatment adherence | Month 9
  A survey to assess dosing of antiretroviral medication

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation for Professional Development, East London, South Africa